CLINICAL TRIAL: NCT00257712
Title: GHRH: Cognition in Aging and MCI
Brief Title: SMART: Somatotrophics, Memory, and Aging Research Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Michael Vitiello, PhD, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 28287-K; R01AG025515 (NIH); R01AG025525-01A1 (NIH)
Record Dates: First submitted 2005-11-21; First posted 2005-11-23 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Aging; Mild Cognitive Impairment
Keywords: Alzheimer's disease; cognition disorders
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Cognition Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: TH9507 human growth hormone releasing hormone (GHRH)
- 2 (Placebo Comparator)
  Interventions: Drug: TH9507 human growth hormone releasing hormone (GHRH)

INTERVENTIONS:
Drug: TH9507 human growth hormone releasing hormone (GHRH) — 1mg subcutaneous injection given daily for 20 weeks

SUMMARY:
The purpose of the SMART study was to better understand whether the body's own production of growth hormone (GH) would improve memory and problem solving ability, or cognitive function. The study was a double blind, placebo-controlled study of the cognitive effects of growth hormone releasing hormone (GHRH) in healthy older men and women and in those with mild cognitive impairment (MCI).

DETAILED DESCRIPTION:
There is considerable and compelling evidence from both the animal and human literature that the actions of the somatotrophic hormonal axis (growth hormone releasing hormone/growth hormone/insulin-like growth factor I) have significant and predictable effects on cognitive function (memory and reasoning ability). A preliminary study has recently shown that five months of growth hormone releasing hormone (GHRH) treatment improves cognitive function in healthy older men and women; there is also preliminary evidence that supports the likelihood of a similar effect in individuals diagnosed with MCI.

The study sample will include 160 adults, ages 55-90, half of whom will be cognitively healthy normal adults and half of whom will meet diagnostic criteria for Mild Cognitive Impairment (MCI). Each of these groups will contain equal numbers of men and women. The treatment with GHRH will be twenty weeks in duration. In light of the documented interactions between estrogens and GHRH/GH/IGF-I, each of the two study arms will contain equal proportions of women not on estrogen replacement therapy (NERT) and women on oral estrogen replacement therapy (ERT). ERT women will maintain a regular steady dosage of estrogens for at least seven days preceding each assessment

Cognitive assessments to evaluate treatment-related changes in memory and thinking abilities, as well as blood collection to evaluate several biomarkers of interest, will be performed at baseline, 10 and 20 weeks of treatment, and ten weeks post-treatment. In addition there will be five medication and symptom monitoring visits during the treatment period.

The study hypotheses are:

H1: Healthy, cognitively normal older men and women treated with GHRH will show beneficial effects in cognitive function, including measures of memory, relative to placebo treated subjects.

H2: MCI patients treated with GHRH will show beneficial effects in cognitive function, including measures of memory, relative to placebo treated MCI patients.

H3: Changes in insulin-like-growth factor (IGF-I) will predict changes in cognition both for normal older adults and for MCI patients treated with GHRH.

ELIGIBILITY:
Inclusion Criteria:

* Able to give and understand informed consent
* Able to communicate in English
* No exclusionary criteria apply
* Age between 55 and 90 years
* Independent in their daily living abilities
* Living at home with a reliable spouse, significant other or caregiver
* Normal PSA (for men) or mammogram (for women) within one year of study entry

The following inclusion criteria will be applied to identify potential MCI participants:

* Memory complaint that can be corroborated by a study partner
* Memory test scores meeting the diagnostic criteria for MCI
* MMSE score greater than 20

The following inclusion criteria will be applied to identify potential normal control participants:

* Cognitive testing does not indicate MCI
* MMSE score greater than 28

Exclusion Criteria:

* Use of medications known to affect the GHRH/GH/IGF-I axis, including transdermal estrogens (use of oral estrogens is not contraindicated)
* Significant medical illness or organ failure, such as uncontrolled hypertension, diabetes, cardiac disease, cerebrovascular disease, chronic obstructive pulmonary disease, kidney and liver disease
* Significant neurologic disease that might affect cognition, such as Alzheimer's disease, stroke, Parkinson's disease, multiple sclerosis, severe head injury with loss of consciousness for more than 30 minutes or with permanent neurologic sequelae
* Personal or strong family history of cancer (especially colon, breast or melanoma)
* Evidence for pituitary disease by history or physical examination
* Symptoms or history of carpal tunnel or a positive Phalen's Test
* Active arthritis
* Significant current psychiatric illness, such as depression, schizophrenia or an Axis II diagnosis suggestive of an inability to successfully complete the study protocol
* Current use of an anti-psychotic, anti-depressant, anti-convulsant, anti-coagulant, anxiolytic or sedative
* Current or planned use of DHEA, testosterone or cognition-enhancing medication (e.g., cholinesterase inhibitors, memantine)
* Weight greater than 150% ideal body weight
* Tobacco use, excessive alcohol intake (more than 2 drinks per day), excessive caffeine intake (more than 4 cups of coffee per day)
* Baseline IGF-I level greater than the mid-range for healthy young adults (250 ng/ml)
* Meets NINCDS/ADRDA criteria for AD

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2006-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in declarative memory, including total recall scores on three tests of memory and on dual task response time (RT), a test of executive function. | Baseline, 10, 20, and 30 weeks

SECONDARY OUTCOMES:
Changes in other areas of cognitive function, including other tests of executive function, tests of lexical access, and tests of cognitive and perceptual-motor processing speed. | Baseline, 10, 20, and 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael V. Vitiello, PhD, Principal Investigator — University of Washington; Suzanne Barsness, RN,MSN,CCRC, Study Director — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Merriam GR, Schwartz RS, Vitiello MV. Growth hormone-releasing hormone and growth hormone secretagogues in normal aging. Endocrine. 2003 Oct;22(1):41-8. doi: 10.1385/ENDO:22:1:41. PMID 14610297
- [Background] Vitiello MV, Moe KE, Merriam GR, Mazzoni G, Buchner DH, Schwartz RS. Growth hormone releasing hormone improves the cognition of healthy older adults. Neurobiol Aging. 2006 Feb;27(2):318-23. doi: 10.1016/j.neurobiolaging.2005.01.010. Epub 2005 Mar 23. PMID 16399214
- [Derived] Friedman SD, Baker LD, Borson S, Jensen JE, Barsness SM, Craft S, Merriam GR, Otto RK, Novotny EJ, Vitiello MV. Growth hormone-releasing hormone effects on brain gamma-aminobutyric acid levels in mild cognitive impairment and healthy aging. JAMA Neurol. 2013 Jul;70(7):883-90. doi: 10.1001/jamaneurol.2013.1425. PMID 23689947
- [Derived] Baker LD, Barsness SM, Borson S, Merriam GR, Friedman SD, Craft S, Vitiello MV. Effects of growth hormone-releasing hormone on cognitive function in adults with mild cognitive impairment and healthy older adults: results of a controlled trial. Arch Neurol. 2012 Nov;69(11):1420-9. doi: 10.1001/archneurol.2012.1970. PMID 22869065